CLINICAL TRIAL: NCT02506608
Title: Natural Sensory Feedback for Phantom Limb Modulation and Therapy
Brief Title: Use of Hand Prosthesis With Direct Nerve Stimulation for Treatment of Phantom Limb Pain
Acronym: EPIONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paolo Maria Rossini (Other)
Collaborators: Aalborg University Hospital (Other); Aalborg University (Other); University of Lausanne Hospitals (Other); University of Freiburg (Other); Université Montpellier (Other); Lund University (Other); Indiana University School of Medicine (Other); Novosense AB (Industry); Mxm-Obelia (Industry); Ecole Polytechnique Fédérale de Lausanne (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor-Investigator, Paolo Maria Rossini, MD, PhD, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIONE-602547-6; no. 602547 (Other Grant/Funding Number: no. 602547)
Record Dates: First submitted 2015-07-20; First posted 2015-07-23 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Phantom Limb Pain
Keywords: Neuroplasticty, Sensory Feedback
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Operation of sensorized hand prosthesis (Experimental): A system composed by the integration of the following non-CE marked medical devices specifically designed for the study will be used in amputees:
  * STIMEP (multichannel electrical stimulator for the peripheral nervous system; AXONIC)
  * TIME 4H Intraneural Electrodes (ALBERT-LUDWIGS-UNIVERSITAET FREIBURG)
  * Sensorized hand Prosthetics for amputees IH2 Prosthetic Azurra Prensilia (Prensilia Ltd.)
  * Prosthetics sensorized hand for amputees DLR / HIT Hand II (Wessling Robotics)
  * ODROID software integration within the afferent and efferent bi-directional control of the robotic hand
  Interventions: Procedure: Operation of sensorized hand prosthesis

INTERVENTIONS:
Procedure: Operation of sensorized hand prosthesis — Four TIME-4H electrodes will be implanted in the median and ulnar of the amputees. The electrodes will be connected with the STIMEP electrical multichannel stimulator. The stimulator will be connected with one of the sensorized prostheses. Afferent and efferent signals will be elaborated and integrated by the ODROID software.
  The amputees will be able to control the prostheses movement and receive a sensory feedback from the prosthesis sensors.
  The use of the prosthesis during different tasks will be considered the intervention.

SUMMARY:
Phantom limb pain (PLP) is a frequent consequence of amputation, and it is notoriously difficult to treat. Amputation usually follows traumatic injuries or surgery following vascular diseases, diabetes, osteomyelitis or tumours in cases where the loss of the limb is required for the survival of the patient. The loss of a limb or other body parts is usually followed by the sensation that the lost body part is still present and can be felt. These phenomena are called, respectively, phantom awareness and phantom sensation. In 50-80% of amputees neuropathic pain develops in the lost limb also referred to as phantom limb pain (PLP). PLP can be related to a certain position or movement of the phantom limb, and might be elicited or worsened by a range of physical factors (e.g. changes in the weather or pressure on the residual limb) and psychological factors (e.g. emotional stress). It is well known that most treatments available for PLP today, such as pharmacological, surgical, anaesthetic, psychological and other, are ineffective. Today it is believed that phantom limb pain may be related to changes in the cortex of the brain. There is evidence that these changes may be modulated - or even reversed - by providing sensory input to the stump or amputation zone. For example, cortical reorganization and alleviation of phantom limb pain has been observed in amputees following intense use of a hand prosthesis. However, there is no consistent knowledge on which type of peripheral sensory feedback may be effective in affecting the cortical plasticity or on how to best apply the sensory feedback. The aim of the proposed research is to create natural, meaningful sensations through providing sensory feedback (i.e. surface or neural electrical stimulation) and the effectiveness to alleviate phantom limb pain and restore the cortical neuroplastic changes.

ELIGIBILITY:
Inclusion Criteria:

* Uni-lateral amputation below the shoulder level
* Other treatments for phantom limb pain should have been tried with poor results
* The subject should experience phantom limb pain at a level of 6 or higher measured on on a visual analog scale (VAS) ranging from 0-10
* Phantom limb pain should be experienced at leaste once a week
* The subject should be in a chronica and stable phase, and the stump should have healed
* The subject should otherwise be healthy and able to carry out the experiment
* If pain medication is used it will be acceptable that the person continues to use the medication

Exclusion Criteria:

* Cognitive impairment
* Pregnancy
* Prior or current psychological diseases such as borderline, schizophrenia, depression or maniodepression
* Acquired brain injury with residual impairment
* Prior neurological or muscoloskeletal diseases
* History of or active substance abuse disorder
* Excessive sensitivity to electrical stimulation with surface electrodes
* Persons with fear for electrical stimulation, pain cannot participate
* Persons that are hypersensitive to electrical stimulation and experience the stimulation as unpleasent cannot participate
* Since the protocol includes MRI scanning of the brain, persons that may feel claustrophobic cannot participate
* Since the protocol includes MRI scanning of the brain, persons that have metal parts in the body (such as pacemakers or bone-screws) cannot participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Phantom limb pain | Change in Phantom Limb Pain daily during the whole study (maximum 1 year per patient)
  Questionnaires (Visual Analogic Scale, Neuropathic Pain Symptom Inventory )
Cortical reorganization | Change in Cortical reorganization before and at the end of 1 year of treatment
  Electroencephalography; Transcranial Magnetic Stimulation and electroencephalography; functional Magnetic Resonance Imaging; Transcranial Magnetic Stimulation ; Somatosensory Evoked Potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Maria Rossini, Roma, IT, Italy